CLINICAL TRIAL: NCT03045900
Title: Measurements of Color Matching and Blending Effect of Translucent and Shaded Bulk-fill Resin Composites [Ex-vivo and In-vivo Study]
Brief Title: Measurements of Color Matching and Blending Effect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abd Allah Nagy Mohamed Abd El Fatah, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-1-3
Record Dates: First submitted 2017-01-31; First posted 2017-02-08 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Translucent bulk-fill resin composite (Active Comparator): *Shaded bulk-fill resin composite. Bulk-fill resin composite which has no shade and could match any other shade. It will be compared for shade accuracy to the haded bulk-fill resin composite.
  Interventions: Other: Shaded bulk-fill resin composite
- Shaded bulk-fill resin composite (Experimental): *Translucent bulk-fill resin composite Bulk-fill resin composite which has a specific shade and should only be filled in teeth with the corresponding shade
  Interventions: Other: Shaded bulk-fill resin composite

INTERVENTIONS:
Other: Shaded bulk-fill resin composite — Dental bulk-fill resin composite with shades A1, A2, A3

SUMMARY:
There is a deficiency in literature which compares the blending effect and color matching of translucent shade bulk-fill resin composite with shaded bulk-fill resin composite. So in this research color matching and blending effect will be instrumentally measured the by a spectrophotometer. A visual assessment also will be done in-vivo and ex-vivo.

DETAILED DESCRIPTION:
Color matching may be the only parameter of treatment with which the patient is concerned. Failure to match the proper color of the teeth may lead to failure of mechanically and biologically successful restoration. Up to 80% of the patients expressed their dissatisfaction with the perceived color of their dental restorations. Thus, proper color reproduction is considered to be one of the most complex and frustrating problems in restorative dentistry.

Polymerisation shrinkage is another serious problem that causes entrapment of stresses that may shorten the clinical life of the restoration. In an effort to reduce this, resin composite is placed in increments as each increment compensate for the previous one. These increments are usually 2 mm each to allow the penetration of curing light. As the resin shade is darker and the filler size is larger, the curing depth will be more limited. So no doubt that the more translucent is the shade of the resin, the higher is the depth of cure. It is noted that, incremental placement is a tedious, time consuming and a very sensitive technique. Improper placement may result in air bubble entrapment or porosity that may result in a weak restoration.

The bulk-fill resin composites specifically designed for large posterior restorations. They represent a new era in direct filling technology and a paradigm shift away from the traditional 2 mm increment system. Bulk-fill resin composite are possible to be cured in a depth of 3.5 to 5.5 mm. This reduces effort and time of the procedure and guarantees a solution for the polymerization shrinkage problem. It is important to note that bulk-fill materials do not constitute a uniform class of materials, they have different consistencies sculptable and flowable. Also some companies produce a translucent shade that should match almost all teeth color as they claim. This is called blending effect where the material can take the shade of the surrounding tooth structure and thus guarantee a solution for color matching problem.

Also there is a deficiency in literature that compares the blending effect and color matching of translucent shade bulk-fill resin composite with shaded bulk-fill resin composite. So in this research we will assess the effect of shaded bulk-fill resin composites against the translucent shade bulk-fill resin composite in-vivo and ex-vivo by spectrophotometer and visual inspection.

ELIGIBILITY:
Inclusion Criteria:

* People with simple class I posterior teeth would be selected without any preference of age or gender.
* Selected molars should only shaded A2, and A3 as these are shades under investigation.
* Patients with multiple caries teeth are preferred.
* Patients should be medically free and with good health.
* Selected molars should be vital.
* Patients should accept participation in the study.

Exclusion Criteria:

* Very deep carious molars that are indicated for root canal treatment or pulp capping.
* Teeth which are cracked, badly decayed crowns, non-restorable, periodontally affected, non-vital or abscessed.
* Patients who refuse to accept participation or had psychological disturbance will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2017-08-15 (Estimated); Study Completion 2017-10-15 (Estimated)

PRIMARY OUTCOMES:
In-vivo visual color matching and blending effect by visual Score from 1 to 5 | Immediately in the same visit
  Visual score from 1-5. The rank (1) is for mismatch or totally unaccepted, (2) is for poor match or hardly accepted, (3) is for good match or accepted, (4) is for close match or small difference, (5) is for exact match or no color difference

IPD SHARING:
Plan to Share IPD: Undecided